CLINICAL TRIAL: NCT03250052
Title: A Phase I Clinical Trial to Evaluate Pharmacokinetic Interactions and Safety Between Fimasartan and Linagliptin in Healthy Male Volunteers
Brief Title: A Clinical Trial to Evaluate Pharmacokinetic Interactions and Safety Between Fimasartan and Linagliptin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BR-FLC-CT-101
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Period 1(fimasartan) x 7days - Period 2(fimasartan + linagliptin) x 7days
  Interventions: Drug: (fimasartan or linagliptin) x 7days; Drug: (fimasartan and linagliptin) x 7days
- Part B (Experimental): Period 1(linagliptin) x 7days - Period 2(fimasartan + linagliptin) x 7days
  Interventions: Drug: (fimasartan or linagliptin) x 7days; Drug: (fimasartan and linagliptin) x 7days

INTERVENTIONS:
Drug: (fimasartan or linagliptin) x 7days — Part A: fimasartan, Part B: linagliptin
Drug: (fimasartan and linagliptin) x 7days — Part A & Part B: Co-administration of fimasartan and linagliptin

SUMMARY:
The purpose of this study is to evaluate pharmacokinetic interactions and safety between fimasartan and linagliptin in healthy male volunteers.

DETAILED DESCRIPTION:
This is an open-label, randomized, multiple-dose, two-period and single-sequence study to evaluate the pharmacokinetics and safety.

ELIGIBILITY:
1. Inclusion Criteria (Total: 5):

1. 19-50 year-old healthy male.
2. 18.5kg/m2 ≤ Body mass index(BMI) ≤ 27kg/m2
3. Subject who has no clinically significant medical history.
4. Subject whose informed consent is obtained and who is willing to comply with protocol.

2. Exclusion Criteria (Total: 19):

1. Sitting systolic blood pressure(SiSBP) ≥ 140mmHg or < 115mmHg / Sitting Diastolic blood pressure(SiDBP) ≥ 90mmHg or < 70mmHg
2. Upper Limits of Normal x 1.5 < Aspartate transaminase(AST), Alanine transminase(ALT), Total bilirubin
3. Creatinine clearance(CrCl) < 80mL/min (using Cockcroft-Gault formula)
4. Positive results in HBsAg, Hepatitis C virus(HCV) Ab, HIV Ag/Ab, Venereal disease research laboratory(VDRL)
5. Participate in another clinical trial within 12 weeks prior to the first administration of Investigational product(IP).

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
[Part A] AUC of fimasartan | 0~24 hour after drug administration
  [Part A] Area under the curve(AUC) of fimasartan in steady state
[Part A] Cmax of fimasartan | 0~24 hour after drug administration
  [Part A] Cmax of fimasartan in steady state
[Part B] AUC of Linagliptin | 0~24 hour after drug administration
  [Part B] Area under the curve(AUC) of Linagliptin in Steady State
[Part B] Cmax of linagliptin | 0~24 hour after drug administration
  [Part B] Cmax of linagliptin in steady state

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, PhD, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang WY, Lee HW, Gwon MR, Cho S, Shim WS, Lee KT, Yang DH, Seong SJ, Yoon YR. A Pharmacokinetic Drug Interaction Between Fimasartan and Linagliptin in Healthy Volunteers. Drug Des Devel Ther. 2020 May 26;14:2101-2111. doi: 10.2147/DDDT.S248205. eCollection 2020. PMID 32546973